CLINICAL TRIAL: NCT01650324
Title: A Double-blind, Randomized, Placebo-controlled, Dose-ranging, Single-dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of DBPR108 in Healthy Male Subjects
Brief Title: A Single-dose Phase 1 Study of DBPR108 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: DBPR108-101
Record Dates: First submitted 2012-07-19; First posted 2012-07-26 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: DBPR108; DPP4; Diabetes; GLP-1; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — DBPR108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DBPR108 (Experimental)
  Interventions: Drug: DBPR108
- matching placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: DBPR108 — DBPR108 capsules in four doses beginning at 25 mg and rising to 600 mg.
  Arms: DBPR108
Drug: matching placebo — Matching placebo capsules in four doses beginning at 25 mg and rising to 600 mg.
  Arms: matching placebo

SUMMARY:
The study is being performed to assess the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) properties of single oral doses of DBPR108 in healthy male subjects.

DETAILED DESCRIPTION:
This study represents the first administration of dipeptidyl peptidase 4 (DPP4) inhibitor DBPR108 to humans to evaluate the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) properties following single oral doses in healthy subjects.

DPP4 is a validated drug target for the treatment of human type 2 diabetes. Objectives of the study will be to characterize the safety and tolerability of single doses of DBPR108; to characterize the single dose PK of DBPR108 in plasma and urine; to characterize the single dose PD of DBPR108 on glucose, glucagon, dipeptidyl peptidase 4 activity, and total and active forms of glucagon-like peptide-1 (GLP-1) in plasma levels and insulin and C-peptide in serum levels.

ELIGIBILITY:
Inclusion Criteria:

* Male with suitable veins for cannulation or repeated venipuncture, and must be able to swallow the study drug intact;
* Aged between 20 and 45 years (inclusive) at the screening visit; and
* Able to provide written informed consent and willing to comply with the study protocol procedures and restrictions.

Exclusion Criteria:

* Has a body weight less than 50 kg and/or body mass index (BMI) less than 18 kg/m2 or greater than 30 kg/m2 at the screening visit;
* Has a creatinine clearance (Ccr) less than 80 mL/min at screening;
* Is not in good general health as judged by the Investigator based on routine medical history, vital signs, physical examination, ECG, laboratory tests, and urinalysis at the screening visit or at admission for the residential period;
* Is not normoglycemic defined as fasting glucose at less than 70 mg/dL (3.9 mmol/L) and greater than 100 mg/dL (5.5 mmol/L);
* Has a platelet count less than 150,000/µL;
* Uses any antihyperglycemic agents at screening or at admission for the residential period;
* Has a history or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs at the screening visit or at admission for the residential period;
* Has a clinically significant psychiatric, renal, hepatic, cardiovascular, gastrointestinal, or neurologic disease at screening or at admission for the residential period;
* Is a smoker and/or has used nicotine-containing products within the last 6 months prior to the screening for the current study and/or has a history of alcohol abuse;
* Has donated blood or participated in another clinical study within 8 weeks preceding the day of admission;
* Excessive intake of caffeine-containing drinks or food (ie, coffee, tea, chocolate, PAOLYTA B Liq, WHISBIH Liq, or cola [more than 6 units of caffeine per day]);
* Use of drugs with enzyme-inducing properties such as St. John's Wort within 4 weeks prior to the first administration of investigational product;
* Has used prescription or nonprescription medication (except for occasional use of paracetamol or nasal spray) or herbal remedies or vitamins or minerals within 2 weeks or 5 half-lives of the drug, whichever is longer, prior to dosing until end of study;
* Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of investigational product;
* Male subjects who are unwilling to use barrier contraception in addition to having their partner use another method of contraception, for the duration of the study and for 3 months after dosing;
* Has a positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV);
* Has received a blood transfusion and/or has HCV infection;
* Positive result on screening for drugs of abuse, alcohol, or cotinine (nicotine) at screening or admission; or
* Involved in the planning or conduct of the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Wanfang Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received either a single oral dose of matching placebo to DBPR108 25 mg, 100 mg, 300 mg, or 600 mg
- DBPR108 25 mg: Participants received a single oral dose of DBPR108 25 mg
- DBPR108 100 mg: Participants received a single oral dose of DBPR108 100 mg
- DBPR108 300 mg: Participants received a single oral dose of DBPR108 300 mg
- DBPR108 600 mg: Participants received a single oral dose of DBPR108 600 mg
Period: Overall Study
Arm/Group | Placebo | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (8) | 26 (2) | 24 (2) | 27 (5) | 26 (6) | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: There were 4 mild adverse events observed during the course of study.
Time Frame: Adverse events were collected from Day -1 (baseline) through the end of the study, up to Day 7.
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Placebo | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 1 | 2

2. Secondary Outcome: Profile of Pharmacokinetics - Area Under the Plasma Concentration-Time Curve (AUC From 0 to Infinity)
Description: Plasma samples were used to determine the AUC from time 0 to infinity for DBPR108. The placebo group is not included in the table below; this outcome measure only evaluated the DBPR108 groups.
Time Frame: predose (0 hr), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post dose
Population: All participants who received a single dose of DBPR108 25 mg, 100 mg, 300 mg, or 600 mg.
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*h/mL | 236 (66.9) | 1310 (290) | 3910 (1200) | 10500 (2400)

3. Secondary Outcome: Profile of Pharmacokinetics - Observed Maximum Plasma Concentration (Cmax)
Description: Plasma samples were used to determine the Cmax for DBPR108. The placebo group is not included in the table below; this outcome measure only evaluated the DBPR108 groups.
Time Frame: predose (0 hr), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post dose
Population: All participants who received a single dose of DBPR108 25 mg, 100 mg, 300 mg, or 600 mg.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 47.2 (23.8) | 187 (33.3) | 571 (158) | 1370 (235)

4. Secondary Outcome: Profile of Pharmacokinetics - Time of Maximum Plasma Concentration (Tmax)
Description: Plasma samples were used to determine the Time of Maximum Plasma Concentration for DBPR108. The placebo group is not included in the table below; this outcome measure only evaluated the DBPR108 groups.
Time Frame: predose (0 hr), 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36 and 48 hrs post dose
Population: All participants who received a single dose of DBPR108 25 mg, 100 mg, 300 mg, or 600 mg.
Measure: Median (Full Range); unit: hrs
Arm/Group | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hrs | 1.50 [1.50 to 4.00] | 4.02 [1.50 to 4.03] | 4.00 [1.00 to 6.00] | 4.01 [2.00 to 6.00]

5. Secondary Outcome: Change of Dipeptidyl Peptidase 4 (DPP4) Activities Between 48 Hrs Post Dose and 0 hr Predose
Description: Change of plasma DPP4 activity at 48 hrs post dose from predose (0 hr). The values were computed as areas under the DPP4 activity-time curve using ANCOVA model, in which the unit of the activity is pmol/min.
Time Frame: predose (0 hr) and 48 hrs post dose
Population: All enrolled participants.
Measure: Geometric Mean (Standard Deviation); unit: h*pmol/min
Groups:
- Placebo: Participants received a single oral dose of matching placebo to DBPR108 25 mg, 100 mg, 300 mg or 600 mg.
Arm/Group | Placebo | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
h*pmol/min | -114 (371) | -925 (464) | -1510 (556) | -2170 (458) | -2350 (671)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day -1 (baseline) through the end of the study, up to Day 7.
Description: No text entered.
Arm/Group | Placebo | DBPR108 25 mg | DBPR108 100 mg | DBPR108 300 mg | DBPR108 600 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | DBPR108 25 mg (N=6) | DBPR108 100 mg (N=6) | DBPR108 300 mg (N=6) | DBPR108 600 mg (N=6)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Platelet Count Decreased
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Infection
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ligament Sprain
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Haematuria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days